CLINICAL TRIAL: NCT06491745
Title: Is Adding Extracorporeal Shock Wave Therapy to Physiotherapy and Corticosteroid Injection Beneficial for Frozen Shoulder?
Brief Title: Is Adding Extracorporeal Shock Wave Therapy to Physiotherapy and Corticosteroid Injection Beneficial for Frozen Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Study Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20231204R; NSTC 113-2314-B-341-003 - (Other Grant/Funding Number: National Science and Technology Council); NSTC 114-2314-B-341-001 - (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Frozen Shoulder; Corticosteroid Injection; Physical Therapy; Extracorporeal Shock Wave Therapy; Rehabilitation
Keywords: Frozen shoulder; corticosteroid injection; physical therapy; extracorporeal shock wave therapy; rehabilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT+PT+corticosteroid injection, ESWT group (Active Comparator): ESWT group. Patients in the ESWT group will receive ESWT, physical therapy, and both shoulder joint (glenohumeral joint, GHJ) and SASD bursa injection for 2 times in a 2-week interval. 3ml triamcinolone (1ml triamcinolone= 10mg) will be added to 3ml 1% xylocaine to make 6ml injectate. Among them, 4ml injectate will be injected into the posterior GHJ with a 7 cm 23-gauge needle under ultrasound (US) guidance. After withdrawing the needle to subcutaneous layer, another 2ml injectate will be injected into the SASD bursa of the affected shoulder under US guidance.
  Interventions: Other: Sham ESWT+PT+corticosteroid injection, SHAM group.
- Sham ESWT+PT+corticosteroid injection, SHAM group. (Active Comparator): SHAM group. The participants will receive the same dosage and technique of corticosteroid posterior GHJ and SASD bursa injection for 2 times at 2 weekly interval as participants do in the ESWT group. For creating a single-blinded condition, they will also receive 4 ESWT treatments at weekly interval except that the energy flux density is set at 0.04 mJ/mm2. For sham ESWT, the machine still makes a noise with every shock wave delivered in order to enhance the sham design.
  Interventions: Other: ESWT+PT+corticosteroid injection, ESWT group

INTERVENTIONS:
Other: ESWT+PT+corticosteroid injection, ESWT group — ESWT group. Patients in the ESWT group will receive ESWT, physical therapy, and both shoulder joint (glenohumeral joint, GHJ) and SASD bursa injection for 2 times in a 2-week interval. 3ml triamcinolone (1ml triamcinolone= 10mg) will be added to 3ml 1% xylocaine to make 6ml injectate. Among them, 4ml injectate will be injected into the posterior GHJ with a 7 cm 23-gauge needle under ultrasound (US) guidance. After withdrawing the needle to subcutaneous layer, another 2ml injectate will be injected into the SASD bursa of the affected shoulder under US guidance.
  Arms: Sham ESWT+PT+corticosteroid injection, SHAM group.
Other: Sham ESWT+PT+corticosteroid injection, SHAM group. — SHAM group. The participants will receive the same dosage and technique of corticosteroid posterior GHJ and SASD bursa injection for 2 times at 2 weekly interval as participants do in the ESWT group. For creating a single-blinded condition, they will also receive 4 ESWT treatments at weekly interval except that the energy flux density is set at 0.04 mJ/mm2. For sham ESWT, the machine still makes a noise with every shock wave delivered in order to enhance the sham design.
  Arms: ESWT+PT+corticosteroid injection, ESWT group

SUMMARY:
Frozen shoulder, or adhesive capsulitis of the shoulder, is a common clinical problem characterized by pain, loss of both passive and active range of motion (ROM) of glenohumeral joint (GHJ), leads to functional limitation, and reduces quality of life. Primary frozen shoulder occurs without any obvious connection to any other condition, and secondary frozen shoulder is related to some medical problems, such as an injury, inflammatory, immunological, and endocrine conditions, or surgery of the shoulder. The prevalence of frozen shoulder is 2%-5% in general population, usually between 40 to 60 years old, and more in female. Diabetes patients have more chance of developing frozen shoulder than general population and the prevalence was 13.4%.

Frozen shoulder is clinically divided into 3 overlapping phases. The painful freezing phase has a duration of 10 to 36 weeks and is characterized by pain and stiffness around the shoulder, which may worsen at night. The frozen phase is characterized by restricted ROM with a gradual relief of pain, which occurs at 4 to 12 months. The thawing phase with spontaneous improvement in the ROM takes 12 to 42 months. .Although frozen shoulder is a self-limited condition, the recovery may be slow and incomplete.

Treatment of frozen shoulder consists of physiotherapy, oral medication (nonsteroidal anti-inflammatory drugs or corticosteroid), intra-articular corticosteroid injection, hydrodilatation, suprascapular nerve block, mobilization, manipulation under anesthesia, and operative intervention (arthroscopic release or open release). Because of the uncertainty of the efficacy and risk of surgical treatment, nonsurgical treatments are more likely chosen by patients. Among them, intra-articular steroid injection and physical therapy are commonly used nonsurgical treatments and have shown some benefits. .Because the clinical picture of frozen shoulder may be similar to, or combining with chronic subacromial bursitis, especially in the freezing stage, concomitant subacromial/subdeltoid (SASD) bursa injection may be needed for treatment of frozen shoulder. In addition, the 3 stages of frozen shoulder often overlap and the clinical symptoms of patients are complex, adjuvant therapy is often needed throughout the course of treatment. Even after physical therapy (PT) and corticosteroid injection, mild to moderate contracture, especially external rotation, abduction, and internal rotation may still be present.

Over the past few years new evidence has emerged on the effectiveness of extracorporeal shock wave therapy (ESWT) in the treatment of many musculoskeletal disorders. Briefly, ESWT has been shown to promote neovasculization, amplify growth factor and protein synthesis, increase of pain inhibiting substance, alteration of pain receptor neurotransmission, and intensification of tissue regeneration. Furthermore, ESWT can produce a cavitation effect between tissues, cause intertissue release, promote the separation of adhesion, and release the adhesive tissue. Because of its analgesic, anti-fibrotic, and anti-inflammatory effect, application of ESWT as main treatment or an adjunct to other interventions has been tried. Knoblock et al found that focused ESWT can reduce pain in painful nodules in Dupuytren's disease; in a randomized controlled trial Chen et al showed focused ESWT was superior to oral corticosteroid for frozen shoulder, although oral corticosteroid is not commonly prescribed for patients with frozen shoulder. Vahdatpour compared ESWT with sham ESWT on treatment of frozen shoulder after 40mg triamcinolone intra-articular injection, and found that ESWT group seemed to have positive effects on treatment, and quicker return to daily life. Another two studies investigating application of radial shock wave to patients with frozen shoulder showed improvement of ROM, even for diabetic patients. A systemic review and meta-analysis also showed ESWT seems beneficial to patients with frozen shoulder and could be used as an adjunct therapy to routine treatments. However, the authors mentioned that the quality of the included randomized controlled trials were hampered by significant heterogeneity regarding long-term analgesia and joint ROM.

Because the effect of ESWT against frozen shoulder has not been well established, we aim to investigate whether adding ESWT to corticosteroid injection and routine PT beneficial for patients with frozen shoulder? We hypothesize that ESWT would be a positive adjunctive therapy in the treatment of frozen shoulder.

DETAILED DESCRIPTION:
Intra-articular and subdeltoid bursal corticosteroid injection and physical therapy (PT) are commonly used nonsurgical treatments for frozen shoulder and have shown good benefits. However, because of complex clinical pictures and overlapping stages, even after the above treatments, pain and contracture of affected shoulder may still exist, and adjuvant therapy is often needed throughout the course of treatment. Over the past few years new evidence has emerged on the effectiveness of extracorporeal shock wave therapy (ESWT) in the treatment of many musculoskeletal disorders. Because of its analgesic, anti-fibrotic effect, and anti-inflammatory effect, application of ESWT to frozen shoulder as an adjunct to other interventions has been tried. However, up to now the effect of ESWT against frozen shoulder has not been well established. We aim to investigate whether adding ESWT to corticosteroid injection and routine PT beneficial for patients with frozen shoulder? This is a prospective single-blind randomized controlled trial. Ninety-four participants with primary frozen shoulder will be recruited from the outpatient clinic of the department of Physical Medicine and Rehabilitation of Shin Kong Wu Ho-Su Memorial Hospital and randomly divided into ESWT group and SHAM group. Each subject in the ESWT group will receive 4 times of ESWT at weekly interval; while participants in the SHAM group receive 4 times of sham ESWT (minimal energy) at weekly interval. Participants in each group also receive 2 times of intraarticular and subdeltoid bursa corticosteroid injection at 2-weekly interval and 8-week physical therapy program.

Outcome measures include the pain visual analog scale (VAS), Shoulder Pain and Disability Index (SPADI), the Shoulder Disability Questionnaire (SDQ), active and passive range of motion (ROM) of the affected shoulder, the 36-item Short Form Health Survey (SF-36), and patient's self evaluation. Evaluations were performed at baseline and at 1, 2, 4, 6 months after the beginning of the treatment. Statistics will be performed after completion of treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 80 years old;
2. shoulder pain for ≥ 1 month;
3. > 30% loss of passive range of motion (ROM) of the affected shoulder in external rotation and/or abduction, comparing with the sound side;
4. pain visual analog scale on maximal passive external rotation or abduction > 4;
5. showing willing to receive ESWT, shoulder joint injection, and attend regular physical therapy programs for 8 weeks.

Exclusion Criteria:

1. severe systemic disorders including cancer, stroke, or cardiopulmonary diseases;
2. uncontrolled DM;
3. rotator cuff tear or calcification of the affected shoulder;
4. fracture, dislocation, or arthritis of the shoulder due to rheumatic disorders;
5. a history of drug allergy to local anesthetics or corticosteroids;
6. pregnancy;
7. receiving ESWT, corticosteroid joint or bursa injection of the affected shoulder during the preceding three months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SPADI is a self-administered questionnaire that evaluate the pain and disability of shoulder diseases. It has 2 subclasses (pain and disability) that consists of 13 items. The pain domain has 5 items and the disabilities domain has 8 items. The SPADI score, which ranges between 0 (best score) and 100 (worst score), is calculated by averaging the scores from the 2 subclasses.

SECONDARY OUTCOMES:
The pain visual analog scale (VAS) | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The pain VAS is obtained using a 100-mm-long horizontal line, with 0 mm on the left, indicating no pain, and 100 mm on the right, indicating very severe pain.22 The pain at rest is defined as rest pain, and pain on maximal abduction of the affected shoulder is defined as activity pain. The reliability of pain VAS is 0.94, but in the absence of a criterion standard for pain, criterion validity cannot be evaluated.

OTHER OUTCOMES:
Range of motion（ROM） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  All the 4 planes of ROM will be measured. It includes abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0° of abduction.
Shoulder Disability Questionnaire（SDQ） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SDQ is a pain-related questionnaire that contains 16 items describing common situations that may induce symptoms in patients with shoulder disorders. The response options are "yes," "no," and "not applicable." The final score is calculated by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst possible condition).
The 36-item Short Form Health Survey（SF-36） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SF-36 is a generic measure of quality of life and is composed of 8 subscales related to the following components: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale generates a score from 0 to 100, and higher scores indicate better health.
Self-assessment of the treatment effect | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=5, effective=4, same=3, worse=2, much worse=1).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan